CLINICAL TRIAL: NCT07065019
Title: Internalized Stigma in Patients With Tooth Loss Due to Periodontitis: A Cross-Sectional Study
Brief Title: Internalized Stigma and Tooth Loss Due to Periodontitis
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Nezahat Arzu Kayar, Principal Investigator, Akdeniz University
Other Study IDs: KAEK-304
Record Dates: First submitted 2025-06-12; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Periodontal Diseases; Tooth Loss
Keywords: periodontal disease; internalized stigma; tooth loss
MeSH Terms: conditions — Periodontal Diseases; Tooth Loss

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stage III periodontitis: The diagnosis of Stage III generalized periodontitis was established based on the presence of one or more of the following clinical and radiographic findings: a probing pocket depth (PD) of ≥ 6 mm and/or clinical attachment loss (CAL) of ≥ 5 mm; radiographic evidence of bone loss extending to the middle or apical third of the root; a history of tooth loss due to periodontitis involving four or fewer teeth; CAL of ≥ 5 mm affecting 30% or more of the dentition; vertical bone loss of ≥ 3 mm; Class II or III furcation involvement; and the presence of moderate ridge defects.
  Interventions: Other: The Internalized Stigma Scale in Mental Illness (ISS)
- Stage IV periodontitis: The diagnosis of Stage IV generalized periodontitis was based on more severe manifestations, including CAL of ≥ 5 mm and radiographic bone loss reaching the middle or apical third of the root. Additionally, patients exhibited tooth loss due to periodontitis affecting five or more teeth, masticatory dysfunction, occlusal dysfunction, severe ridge defects, and/or signs of secondary occlusal trauma.
  Interventions: Other: The Internalized Stigma Scale in Mental Illness (ISS)

INTERVENTIONS:
Other: The Internalized Stigma Scale in Mental Illness (ISS) — The ISS consists of 29 items and is a self-report scale assessing internalized stigma. ISS includes 5 subscales: 1. Alienation (6 items), 2. Confirmation of Stereotypes (7 items), 3. Perceived Discrimination (5 items), 4. Social Withdrawal (6 items), 5. Resistance to Stigmatization (5 items). ISS is a Likert-type scale calculated as 'strongly disagree' (1 point), 'disagree' (2 points), 'agree' (3 points), 'strongly agree' (4 points). The items of the 'Resistance to stigmatization' subscale are reverse scored. High scores on this scale indicate how aggressive the person's internalized stigma is negatively. ISS has been adapted for many diseases other than mental illnesses in our country and its validity and reliability have been demonstrated.

SUMMARY:
Internalized stigma refers to the adoption of negative judgments, beliefs, stereotypes and stigmatizing views imposed by society.

The aim of this study was to investigate internalized stigma in patients with tooth loss due to periodontitis.

This study included a total of 155 volunteer individuals diagnosed with Stage III or Stage IV periodontitis. 'Internalized Stigma Scale in Mental Illness', 'Individual Information Collection Form' including sociodemographic data and 'Patient Evaluation Form' including clinical periodontal parameters were obtained from these volunteers.

DETAILED DESCRIPTION:
This study included 155 volunteer individuals diagnosed with Stage III and Stage IV periodontitis who applied to Akdeniz University Faculty of Dentistry Periodontology Clinic between May 2023 and July 2024. 'Internalized Stigma Scale in Mental Illness', 'Individual Information Collection Form' including sociodemographic data and 'Patient Evaluation Form' including clinical periodontal parameters were obtained from these volunteers. This study was conducted in accordance with the Helsinki Declaration of 1975, as revised in 2013. After the rationale and method of the study were explained to the volunteers included in the study, a minimum informed consent form was signed.

This study included patients diagnosed with Generalized Stage III and Generalized Stage IV periodontitis, according to the criteria defined in the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions.

Data Collection Procedure and Indexes:

The internalized stigma scale(ISS) consists of 29 items and is a self-report scale assessing internalized stigma. ISS includes 5 subscales: 1. Alienation (6 items), 2. Confirmation of Stereotypes (7 items), 3. Perceived Discrimination (5 items), 4. Social Withdrawal (6 items), 5. Resistance to Stigmatization (5 items). ISS is a Likert-type scale calculated as 'strongly disagree' (1 point), 'disagree' (2 points), 'agree' (3 points), 'strongly agree' (4 points). The items of the 'Resistance to stigmatization' subscale are reverse scored. High scores on this scale indicate how aggressive the person's internalized stigma is negatively. ISS has been adapted for many diseases other than mental illnesses in our country and its validity and reliability have been demonstrated.In a recent study . ISS has been shown to be valid and reliable in halitosis (Cronbach's alpha = 0.89). In the current study, the Internalized Stigma of Mental Illness (ISMI) Scale demonstrated high internal consistency, with a Cronbach's alpha coefficient of 0.947.

ELIGIBILITY:
Inclusion Criteria:

* Tooth loss due to interproximal CAL and mobility caused by periodontal disease
* Patients must be over 18 and under 65 years of age
* Demonstrate adequate cognitive function and comprehension skills, as assessed through clinical observation.
* Know how to read and write
* Patients do not have any neurological disease that may affect the perception of internalized stigma
* Patients volunteering to participate in the study

Exclusion Criteria:

* Has any medical condition or neurological disease that may affect the perception of internalized stigma
* Patients with tooth loss due to reasons other than interproximal CAC and mobility caused by periodontal disease
* The appearance of teeth lost due to periodontitis concealed by a fixed or removable prosthesis
* Those who do not want to participate in the survey
* Lack sufficient cognitive and comprehension abilities as determined through clinical observation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study included patients diagnosed with Generalized Stage III and Generalized Stage IV periodontitis, according to the criteria defined in the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions
Sampling Method: Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Internalized stigma in patients with tooth loss due to periodontitis | 6 months
  Tooth loss due to periodontitis refers to the extraction or spontaneous exfoliation of a tooth as a direct consequence of the progressive destruction of the tooth-supporting structures, including the periodontal ligament, alveolar bone, and connective tissue attachment. This destruction results from chronic inflammation and tissue breakdown caused by periodontal pathogens. Teeth are considered lost due to periodontitis when mobility, severe attachment loss, and bone resorption render them non-functional, painful, or unsalvageable despite periodontal therapy.
  Internalized Stigma of Mental Illness Scale assessment was performed in patients with tooth loss due to periodontitis.Internalized Stigma of Mental Illness Scale is a Likert-type scale calculated as 'strongly disagree' (1 point), 'disagree' (2 points), 'agree' (3 points), 'strongly agree' (4 points).High scores on this scale indicate how aggressive the person's internalized stigma is negatively.
The correlation between potential internalized stigma and different sociodemographic factors. | 6 months
  Sociodemographic data such as age, gender, marital status, education level, income level, smoking status, presence of systemic diseases, reason for referral, and frequency of tooth brushing were recorded.Internalized Stigma of Mental Illness Scale is a Likert-type scale calculated as 'strongly disagree' (1 point), 'disagree' (2 points), 'agree' (3 points), 'strongly agree' (4 points).High scores on this scale indicate how aggressive the person's internalized stigma is negatively.

SECONDARY OUTCOMES:
The correlation between potential internalized stigma and plaque index | 6 months
  These measurements were taken at specific sites around each tooth via a Williams periodontal probe.
  The Plaque Index (PI), as described by Silness and Löe, is used to assess the thickness of plaque at the gingival area.Without using disclosing agents, the presence of plaque is assessed visually and by gently passing the probe along the gingival margin. Each surface is scored on a scale from 0 to 3:
  Score 0: No plaque.
  Score 1: A film of plaque adhering to the free gingival margin and adjacent area of the tooth, detectable only by running a probe across the tooth surface.
  Score 2: Moderate accumulation of soft deposits within the gingival pocket or on the tooth and gingival margin, visible to the naked eye.
  Score 3: Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
The correlation between potential internalized stigma and gingival index (GI) | 6 months
  The GI was measured at six sites per tooth, according to Löe & Silness: 0- Normal gingiva; 1- Mild inflammation with slight color change, mild alteration of gingival surface structure and no bleeding on probing; 2- Moderate inflammation with edema, redness, swelling and bleeding on probing; 3- Severe inflammation with marked edema and redness, ulceration and tendency to bleed spontaneously.These measurements were taken at specific sites around each tooth via a graduated periodontal probe.
The correlation between potential internalized stigma and probing pocket depth | 6 months
  Probing pocket depth were taken at six sites/tooth and recorded using a Williams periodontal probe. PPD is measured as the distance from the gingival margin to the base of the gingival sulcus or periodontal pocket. A calibrated periodontal probe is gently inserted parallel to the long axis of the tooth into the sulcus or pocket until slight resistance is felt at the base. The depth is recorded in millimeters at six sites per tooth: mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual. This measurement reflects the current inflammatory status and pocket formation around the tooth.
The correlation between potential internalized stigma and clinical attachment loss | 6 months
  The CAL is measured by determining the distance from the cementoenamel junction (CEJ) to the base of the periodontal pocket or sulcus. A calibrated periodontal probe is gently inserted into the gingival sulcus or pocket, and the probing depth (PD) is recorded. If the gingival margin is located coronal to the CEJ, the distance from the gingival margin to the CEJ is subtracted from the probing depth. If the gingival margin is apical to the CEJ (in cases of recession), this distance is added to the probing depth. The resulting value represents the CAL, which reflects the extent of periodontal support loss.

CONTACTS AND LOCATIONS:
Overall Officials: Nezahat Arzu Kayar, Phd, Principal Investigator — Akdeniz University
Locations (2):
- Turkey (Türkiye) (2):
  - Nezahat Arzu Kayar, Antalya, Antalya
  - Nezahat Arzu Kayar, Konyaalti, Antalya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sum MY, Wong CTW, Chu ST, Li A, Lee AHT, Chen EYH, Chan SKW. Systematic review and meta-analysis of internalised stigma and stigma resistance in patients with psychosis: The impact of individualism-collectivism culture and other individual factors. Int J Soc Psychiatry. 2024 Jun;70(4):639-652. doi: 10.1177/00207640231216924. Epub 2024 Jan 26. PMID 38279534
- [Background] Zain Ul Abideen M, Ali Bushara NA, Nadeem Baig M, Dilshad Siddiqui Y, Ejaz I, Tareen J, Siddiqui AA. Shining a Spotlight on Stigma: Exploring Its Impact on Oral Health-Seeking Behaviours Through the Lenses of Patients and Caregivers. Cureus. 2024 Jun 24;16(6):e63025. doi: 10.7759/cureus.63025. eCollection 2024 Jun. PMID 39050292